CLINICAL TRIAL: NCT06109181
Title: A Phase 1/2 Study of the Safety and Efficacy of LX2020 Gene Therapy in Patients With Arrhythmogenic Cardiomyopathy Due to a Plakophilin-2 Pathogenic Variant
Brief Title: Gene Therapy for ACM Due to a PKP2 Pathogenic Variant
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lexeo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LX2020-01
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Arrhythmogenic Cardiomyopathy; PKP2-ACM; PKP2-ARVC
Keywords: Arrhythmogenic Cardiomyopathy; ACM; Cardiomyopathy; ARVC; Arrhythmogenic Right Ventricular; Arrhythmogenic Right Ventricular Dysplasia; Genetic cardiomyopathy; Gene Therapy; PKP2 Gene; Plakophilin-2; LX2020; HEROIC-PKP2; Ventricular Arrhythmia; PVCs; Sudden Cardiac Death; Cardiac Arrest
MeSH Terms: conditions — Cardiomyopathies; Arrhythmogenic Right Ventricular Dysplasia; Death, Sudden, Cardiac; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LX2020 (Experimental): Single ascending dose of LX2020, with a starting dose of 2.0 x10^13 gc/kg, in multiple cohorts
  Interventions: Genetic: LX2020

INTERVENTIONS:
Genetic: LX2020 — LX2020 is an adeno-associated viral vector encoding the human Plakophilin-2 (PKP2) gene (AAVrh.10hPKP2)

SUMMARY:
This is a Phase 1/2, first-in-human, open-label, intravenous, dose-escalating, multicenter trial that is designed to assess the safety and tolerability of LX2020 in adult patients with PKP2-ACM

ELIGIBILITY:
Selected Inclusion Criteria:

* Adults with a clinical diagnosis of ACM meeting the 2010 revised Task Force Criteria (TFC)
* Genetic testing documenting a pathogenic or likely pathogenic variant in PKP2
* Frequent premature ventricular complexes (PVCs)
* Implantable cardioverter-defibrillator (ICD) implantation ≥ 12 weeks prior to the pre-screening MRI
* Left ventricular ejection fraction ≥ 40%

Selected Exclusion Criteria:

* Evidence of variant(s) in addition to PKP2 that meets the standard criteria to be considered pathogenic or likely pathogenic for ACM
* Other cardiac abnormalities as specified in the protocol
* New York Heart Association Functional Class IV at the time of consent
* History of prior gene transfer therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who experienced at least 1 treatment emergent adverse event (TEAE) and/or 1 treatment emergent serious adverse event (TESAE). | 12 months
  Evaluation of Safety and Tolerability of LX2020

OTHER OUTCOMES:
Selected Exploratory | 12 months
  Change in the frequency of ventricular arrhythmias from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: LEXEO Clinical Trials, Study Director — Lexeo Therapeutics
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Rochester, Rochester, New York
  - Medical University of South Carolina, Charleston, South Carolina